CLINICAL TRIAL: NCT03345420
Title: NOVEMBER (Novem- (9), BrEast Radiation), A Phase II Trial of a 9 Day Course of Whole Breast Radiotherapy for Early Stage Breast Cancer
Brief Title: Hypofractionated Radiation Therapy in Treating Patients With Stage 0-IIB Breast Cancer
Acronym: NOVEMBER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI103976; NCI-2017-02018 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HCI103976 (Other: Huntsman Cancer Institute/University of Utah)
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Ductal Breast Carcinoma In Situ; Invasive Breast Carcinoma; Stage 0 Breast Cancer; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Within 12 weeks after breast conserving surgery, patients undergo hypofractionated radiation therapy for 9 fractions over 2 weeks.
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated Radiotherapy; hypofractionation

SUMMARY:
This phase II trial studies how well hypofractionated radiation therapy works in treating patients with stage 0-IIB breast cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
Adjuvant radiation therapy (RT) plays an important role in successful breast conservation in early-stage breast cancer and has been shown to significantly reduce the risk of breast cancer recurrence over surgery alone. Adding breast radiation to lumpectomy has allowed women to keep their natural breast, as multiple randomized trials have demonstrated equivalent overall and disease-free survival compared to a mastectomy. Meta-analyses have concluded that post-lumpectomy radiation improves breast cancer survival, with an estimated 1 life saved for every 4 recurrences prevented. An important component of radiation therapy is the time-dose-fractionation schedule. Up until the last decade, the standard radiation schedule in North America involved 6-8 weeks of daily radiation.

This study proposes that fractionation will provide a significant improvement in convenience and cost effectiveness, while delivering equivalent cancer control.

This will be a phase II single arm non-inferiority trial. Trial patients will receive 9 fractions hypofractionated radiation. Patients will be evaluated for breast photographic cosmetic scores with hypofractionated radiation compared to standard fractionation 24 months after radiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive carcinoma and/or ductal carcinoma in situ (DCIS) of the breast
* Final pathologic Tis, T1-T3, all must be N0 and M0 status.
* Negative inked histologic margins from lumpectomy, with the exception of a focus of positive margin at the pectoralis fascia
* Radiation oncologist does not plan to treat regional lymph nodes beyond standard whole breast tangent fields
* Lumpectomy with negative lymph node on surgical evaluation (Isolated tumor cells in lymph nodes will be permitted). Patients with invasive carcinoma ≥ 70 yrs and with ER+ positive tumor ≤ 2.0cm may enroll without surgical lymph node evaluation, per section 5.1. Patients with Ductal Carcinoma In Situ (DCIS) of the breast only may enroll without surgical lymph node evaluation.
* Negative serum or urine beta-human chorionic gonadotropin (HCG) in women of child-bearing potential =< 7 days prior to registration

  * A female of childbearing potential is a sexually mature female who has not undergone a hysterectomy or bilateral oophorectomy and has not been naturally postmenopausal for at least 12 consecutive months
* Women of child-bearing potential must agree to utilize a form of birth control or agree to undergo sexual abstinence during radiation therapy
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines

Exclusion Criteria:

* Prior radiation therapy to the chest, neck or axilla
* Prior history of ipsilateral breast cancer (invasive disease or DCIS); lobular carcinoma in situ (LCIS) and benign breast disease is allowed
* History of prior or concurrent contralateral invasive breast cancer; benign breast disease, LCIS or DCIS of contralateral breast is allowed
* Active collagen vascular diseases, such as: systemic lupus erythematous, scleroderma, or dermatomyositis
* Significant post lumpectomy complications requiring an unplanned re-operation or admission for intravenous (IV) antibiotics; re-operation for margins evaluation or nodal evaluation is acceptable
* Co-existing medical conditions with life expectancy < 5 years
* Other malignancy within 5 years of registration with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the cervix
* Neoadjuvant chemotherapy or adjuvant chemotherapy delivered before radiation
* Neuroendocrine carcinoma or sarcoma histology
* Concurrent radiation sensitizing medications concurrent with radiation, per treatment physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2025-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Poppe, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Early Breast Cancer Trialists' Collaborative Group. Effects of radiotherapy and surgery in early breast cancer. An overview of the randomized trials. N Engl J Med. 1995 Nov 30;333(22):1444-55. doi: 10.1056/NEJM199511303332202. PMID 7477144
- [Background] Vinh-Hung V, Verschraegen C. Breast-conserving surgery with or without radiotherapy: pooled-analysis for risks of ipsilateral breast tumor recurrence and mortality. J Natl Cancer Inst. 2004 Jan 21;96(2):115-21. doi: 10.1093/jnci/djh013. PMID 14734701
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] van Dongen JA, Voogd AC, Fentiman IS, Legrand C, Sylvester RJ, Tong D, van der Schueren E, Helle PA, van Zijl K, Bartelink H. Long-term results of a randomized trial comparing breast-conserving therapy with mastectomy: European Organization for Research and Treatment of Cancer 10801 trial. J Natl Cancer Inst. 2000 Jul 19;92(14):1143-50. doi: 10.1093/jnci/92.14.1143. PMID 10904087
- [Background] Veronesi U, Cascinelli N, Mariani L, Greco M, Saccozzi R, Luini A, Aguilar M, Marubini E. Twenty-year follow-up of a randomized study comparing breast-conserving surgery with radical mastectomy for early breast cancer. N Engl J Med. 2002 Oct 17;347(16):1227-32. doi: 10.1056/NEJMoa020989. PMID 12393819
- [Background] Frandsen J, Ly D, Cannon G, Suneja G, Matsen C, Gaffney DK, Wright M, Kokeny KE, Poppe MM. In the Modern Treatment Era, Is Breast Conservation Equivalent to Mastectomy in Women Younger Than 40 Years of Age? A Multi-Institution Study. Int J Radiat Oncol Biol Phys. 2015 Dec 1;93(5):1096-103. doi: 10.1016/j.ijrobp.2015.08.044. Epub 2015 Sep 1. PMID 26581146
- [Background] Owen JR, Ashton A, Bliss JM, Homewood J, Harper C, Hanson J, Haviland J, Bentzen SM, Yarnold JR. Effect of radiotherapy fraction size on tumour control in patients with early-stage breast cancer after local tumour excision: long-term results of a randomised trial. Lancet Oncol. 2006 Jun;7(6):467-71. doi: 10.1016/S1470-2045(06)70699-4. PMID 16750496
- [Background] Haviland JS, Owen JR, Dewar JA, Agrawal RK, Barrett J, Barrett-Lee PJ, Dobbs HJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Simmons S, Sydenham MA, Venables K, Bliss JM, Yarnold JR; START Trialists' Group. The UK Standardisation of Breast Radiotherapy (START) trials of radiotherapy hypofractionation for treatment of early breast cancer: 10-year follow-up results of two randomised controlled trials. Lancet Oncol. 2013 Oct;14(11):1086-1094. doi: 10.1016/S1470-2045(13)70386-3. Epub 2013 Sep 19. PMID 24055415
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Background] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- [Background] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Background] Romestaing P, Lehingue Y, Carrie C, Coquard R, Montbarbon X, Ardiet JM, Mamelle N, Gerard JP. Role of a 10-Gy boost in the conservative treatment of early breast cancer: results of a randomized clinical trial in Lyon, France. J Clin Oncol. 1997 Mar;15(3):963-8. doi: 10.1200/JCO.1997.15.3.963. PMID 9060534
- [Background] Vrieling C, Collette L, Fourquet A, Hoogenraad WJ, Horiot JC, Jager JJ, Pierart M, Poortmans PM, Struikmans H, Van der Hulst M, Van der Schueren E, Bartelink H. The influence of the boost in breast-conserving therapy on cosmetic outcome in the EORTC "boost versus no boost" trial. EORTC Radiotherapy and Breast Cancer Cooperative Groups. European Organization for Research and Treatment of Cancer. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):677-85. doi: 10.1016/s0360-3016(99)00211-4. PMID 10524422
- [Background] Cante D, Franco P, Sciacero P, Girelli G, Pasquino M, Casanova Borca V, Tofani S, Porta MR, Ricardi U. Hypofractionated whole-breast radiotherapy and concomitant boost after breast conservation in elderly patients. Tumori. 2016 Mar-Apr;102(2):196-202. doi: 10.5301/tj.5000402. Epub 2015 Aug 26. PMID 26350199
- [Background] Franco P, Zeverino M, Migliaccio F, Cante D, Sciacero P, Casanova Borca V, Torielli P, Arrichiello C, Girelli G, La Porta MR, Tofani S, Numico G, Ricardi U. Intensity-modulated and hypofractionated simultaneous integrated boost adjuvant breast radiation employing statics ports of tomotherapy (TomoDirect): a prospective phase II trial. J Cancer Res Clin Oncol. 2014 Jan;140(1):167-77. doi: 10.1007/s00432-013-1560-8. Epub 2013 Nov 30. PMID 24292425
- [Background] Ghannam AA, Khedr RA. An accelerated hypofractionated schedule with a daily concomitant boost after breast conservation surgery: the feasibility and toxicity. J Egypt Natl Canc Inst. 2016 Mar;28(1):39-44. doi: 10.1016/j.jnci.2016.01.002. Epub 2016 Jan 28. PMID 26833225
- [Background] Mondal D, Julka PK, Sharma DN, Jana M, Laviraj MA, Deo SV, Roy S, Guleria R, Rath GK. Accelerated hypofractionated adjuvant whole breast radiation with simultaneous integrated boost using volumetric modulated arc therapy for early breast cancer: A phase I/II dosimetric and clinical feasibility study from a tertiary cancer care centre of India. J Egypt Natl Canc Inst. 2017 Mar;29(1):39-45. doi: 10.1016/j.jnci.2017.01.005. PMID 28343538
- [Background] Freedman GM, White JR, Arthur DW, Allen Li X, Vicini FA. Accelerated fractionation with a concurrent boost for early stage breast cancer. Radiother Oncol. 2013 Jan;106(1):15-20. doi: 10.1016/j.radonc.2012.12.001. Epub 2013 Jan 17. PMID 23333014
- [Background] FAST Trialists group; Agrawal RK, Alhasso A, Barrett-Lee PJ, Bliss JM, Bliss P, Bloomfield D, Bowen J, Brunt AM, Donovan E, Emson M, Goodman A, Harnett A, Haviland JS, Kaggwa R, Morden JP, Robinson A, Simmons S, Stewart A, Sydenham MA, Syndikus I, Tremlett J, Tsang Y, Wheatley D, Venables K, Yarnold JR. First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015). Radiother Oncol. 2011 Jul;100(1):93-100. doi: 10.1016/j.radonc.2011.06.026. PMID 21752481
- [Background] Bekelman JE, Sylwestrzak G, Barron J, Liu J, Epstein AJ, Freedman G, Malin J, Emanuel EJ. Uptake and costs of hypofractionated vs conventional whole breast irradiation after breast conserving surgery in the United States, 2008-2013. JAMA. 2014 Dec 17;312(23):2542-50. doi: 10.1001/jama.2014.16616. PMID 25494006
- [Background] Haffty BG, Buchholz TA. Hypofractionated breast radiation: preferred standard of care? Lancet Oncol. 2013 Oct;14(11):1032-1034. doi: 10.1016/S1470-2045(13)70405-4. No abstract available. PMID 24079860
- [Background] Rajagopalan MS, Flickinger JC, Heron DE, Beriwal S. Changing practice patterns for breast cancer radiation therapy with clinical pathways: An analysis of hypofractionation in a large, integrated cancer center network. Pract Radiat Oncol. 2015 Mar-Apr;5(2):63-9. doi: 10.1016/j.prro.2014.10.004. PMID 25748004
- [Background] Wang EH, Mougalian SS, Soulos PR, Rutter CE, Evans SB, Haffty BG, Gross CP, Yu JB. Adoption of hypofractionated whole-breast irradiation for early-stage breast cancer: a National Cancer Data Base analysis. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):993-1000. doi: 10.1016/j.ijrobp.2014.06.038. Epub 2014 Aug 19. PMID 25149661
- [Background] Fowler JF. The linear-quadratic formula and progress in fractionated radiotherapy. Br J Radiol. 1989 Aug;62(740):679-94. doi: 10.1259/0007-1285-62-740-679. No abstract available. PMID 2670032
- [Background] Matthews JH, Meeker BE, Chapman JD. Response of human tumor cell lines in vitro to fractionated irradiation. Int J Radiat Oncol Biol Phys. 1989 Jan;16(1):133-8. doi: 10.1016/0360-3016(89)90020-5. PMID 2912934
- [Background] Steel GG, Deacon JM, Duchesne GM, Horwich A, Kelland LR, Peacock JH. The dose-rate effect in human tumour cells. Radiother Oncol. 1987 Aug;9(4):299-310. doi: 10.1016/s0167-8140(87)80151-2. PMID 3317524
- [Background] Falchook AD, Green R, Knowles ME, Amdur RJ, Mendenhall W, Hayes DN, Grilley-Olson JE, Weiss J, Reeve BB, Mitchell SA, Basch EM, Chera BS. Comparison of Patient- and Practitioner-Reported Toxic Effects Associated With Chemoradiotherapy for Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2016 Jun 1;142(6):517-23. doi: 10.1001/jamaoto.2016.0656. PMID 27149571
- [Background] Kanatas A, Velikova G, Roe B, Horgan K, Ghazali N, Shaw RJ, Rogers SN. Patient-reported outcomes in breast oncology: a review of validated outcome instruments. Tumori. 2012 Nov;98(6):678-88. doi: 10.1177/030089161209800602. PMID 23389352
- [Background] Oberguggenberger A, Hubalek M, Sztankay M, Meraner V, Beer B, Oberacher H, Giesinger J, Kemmler G, Egle D, Gamper EM, Sperner-Unterweger B, Holzner B. Is the toxicity of adjuvant aromatase inhibitor therapy underestimated? Complementary information from patient-reported outcomes (PROs). Breast Cancer Res Treat. 2011 Jul;128(2):553-61. doi: 10.1007/s10549-011-1378-5. Epub 2011 Feb 11. PMID 21311968
- [Background] Koslow S, Pharmer LA, Scott AM, Stempel M, Morrow M, Pusic AL, King TA. Long-term patient-reported satisfaction after contralateral prophylactic mastectomy and implant reconstruction. Ann Surg Oncol. 2013 Oct;20(11):3422-9. doi: 10.1245/s10434-013-3026-2. Epub 2013 May 30. PMID 23720070
- [Background] Rosson GD, Shridharani SM, Magarakis M, Manahan MA, Basdag B, Gilson MM, Pusic AL. Quality of life before reconstructive breast surgery: A preoperative comparison of patients with immediate, delayed, and major revision reconstruction. Microsurgery. 2013 May;33(4):253-8. doi: 10.1002/micr.22081. Epub 2013 Feb 17. PMID 23417854
- [Background] Fuzesi S, Cano SJ, Klassen AF, Atisha D, Pusic AL. Validation of the electronic version of the BREAST-Q in the army of women study. Breast. 2017 Jun;33:44-49. doi: 10.1016/j.breast.2017.02.015. Epub 2017 Mar 7. PMID 28279888
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Olivotto IA, Whelan TJ, Parpia S, Kim DH, Berrang T, Truong PT, Kong I, Cochrane B, Nichol A, Roy I, Germain I, Akra M, Reed M, Fyles A, Trotter T, Perera F, Beckham W, Levine MN, Julian JA. Interim cosmetic and toxicity results from RAPID: a randomized trial of accelerated partial breast irradiation using three-dimensional conformal external beam radiation therapy. J Clin Oncol. 2013 Nov 10;31(32):4038-45. doi: 10.1200/JCO.2013.50.5511. Epub 2013 Jul 8. PMID 23835717
- [Background] Vrieling C, Collette L, Bartelink E, Borger JH, Brenninkmeyer SJ, Horiot JC, Pierart M, Poortmans PM, Struikmans H, Van der Schueren E, Van Dongen JA, Van Limbergen E, Bartelink H. Validation of the methods of cosmetic assessment after breast-conserving therapy in the EORTC "boost versus no boost" trial. EORTC Radiotherapy and Breast Cancer Cooperative Groups. European Organization for Research and Treatment of Cancer. Int J Radiat Oncol Biol Phys. 1999 Oct 1;45(3):667-76. doi: 10.1016/s0360-3016(99)00215-1. PMID 10524421
- [Background] Hughes KS, Schnaper LA, Bellon JR, Cirrincione CT, Berry DA, McCormick B, Muss HB, Smith BL, Hudis CA, Winer EP, Wood WC. Lumpectomy plus tamoxifen with or without irradiation in women age 70 years or older with early breast cancer: long-term follow-up of CALGB 9343. J Clin Oncol. 2013 Jul 1;31(19):2382-7. doi: 10.1200/JCO.2012.45.2615. Epub 2013 May 20. PMID 23690420
- [Background] Mundy LR, Homa K, Klassen AF, Pusic AL, Kerrigan CL. Breast Cancer and Reconstruction: Normative Data for Interpreting the BREAST-Q. Plast Reconstr Surg. 2017 May;139(5):1046e-1055e. doi: 10.1097/PRS.0000000000003241. PMID 28445351
- [Background] National Institute for Health and Care Excellence. Guide to the Methods of Technology Appraisal 2013 [Internet]. London: National Institute for Health and Care Excellence (NICE); 2013 Apr 4. Process and Methods Guides No. 9. Available from http://www.ncbi.nlm.nih.gov/books/NBK395867/ PMID 27905712
- [Result] Poppe MM, Boucher K, Gaffney DK, Brownson KE, Smith G, Howell JN, Ticona FF, Kim J, Burt L, Cannon D, Kokeny K. NOVEMBER, A Phase 2 Trial of a 9-Day Course of Whole Breast Radiation Therapy With a Simultaneous Lumpectomy Boost for Early-Stage Breast Cancer. Int J Radiat Oncol Biol Phys. 2025 Sep 1;123(1):141-149. doi: 10.1016/j.ijrobp.2025.03.078. Epub 2025 May 2. PMID 40314623
- See also: NOVEMBER, A Phase 2 Trial of a 9-Day Course of Whole Breast Radiation Therapy With a Simultaneous Lumpectomy Boost for Early-Stage Breast Cancer — https://pubmed.ncbi.nlm.nih.gov/40314623/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Within 12 weeks after breast conserving surgery, participants undergo hypofractionated radiation therapy for 9 fractions over 2 weeks.
  Hypofractionated Radiation Therapy: Undergo hypofractionated radiation therapy
Period: Overall Study
Arm/Group | Treatment
Started | 102
Hypofractionated Radiotherapy | 102
Completed | 101
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.71 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 92
  More than one race | 0
  Unknown or Not Reported | 3
Breast photographic cosmetic scores [Count of Participants; unit: Participants] — The EORTC (European Organisation for Research and Treatment of Cancer) Breast Cosmetic Rating system is a blinded digital photographic method that compares the radiated breast with the contralateral untreated side and evaluates: Size, shape, location of the areola/nipple, appearance of the surgical scar, skin pigmentation changes, presence of telangiectasia and a global cosmetic score based on all of the factors. Characteristics are graded on a four-point scale: 0, excellent or no difference; 1, good or small difference; 2, fair or moderate difference; and 3, poor or large difference. Population: Of 102 total enrolled participants, images from 89 participants at baseline were available and of sufficient quality to be reviewed and scored by the 3 unbiased reviewers.
  Participants
    Excellent: number analyzed (Participants) | 89
    Excellent | 36
    Good: number analyzed (Participants) | 89
    Good | 32
    Fair: number analyzed (Participants) | 89
    Fair | 19
    Poor: number analyzed (Participants) | 89
    Poor | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants by EORTC Breast Cosmetic Rating Score at 24 Months Post-radiation Therapy
Description: The EORTC (European Organisation for Research and Treatment of Cancer) Breast Cosmetic Rating system is a blinded digital photographic method that compares the radiated breast with the contralateral untreated side and evaluates: Size, shape, location of the areola/nipple, appearance of the surgical scar, skin pigmentation changes, presence of telangiectasia and a global cosmetic score based on all of the factors. Characteristics are graded on a four-point scale: 0, excellent or no difference; 1, good or small difference; 2, fair or moderate difference; and 3, poor or large difference. Images taken at the 24 month timepoint were assessed by 3 unbiased reviewers including a radiation oncologist, surgeon and nurse. The data is presented as the count of participants meeting the overall rating criteria as assessed by these reviewers.
Time Frame: Up to 24 months post radiation therapy (RT)
Population: Of 102 total enrolled participants, images from 78 participants at this timepoint were available and of sufficient quality to be reviewed and scored by the 3 unbiased reviewers.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 78
Participants
  Excellent | 17
  Good | 26
  Fair | 24
  Poor | 11

2. Secondary Outcome: Quality of Life as Measured by Breast-Q Questionnaire Scores at 6 Month Post-RT Timepoint
Description: * Assessed 4 subscales: satisfaction with breasts, psychosocial well-being, physical well-being, and sexual well-being.
  * Score from 0 (worst) to 100 (best). Higher scores reflect a better outcome.
Time Frame: 6 months post RT
Population: * 80 sexual well-being subscale questionnaires were completed at this timepoint
  * 95 satisfaction with breasts subscale questionnaires were completed at this timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 96
score on a scale
  Physical well-being | 68.2 (22.9)
  Psychosocial well-being | 79.6 (20.2)
  Sexual well-being: number analyzed (Participants) | 80
  Sexual well-being | 63.4 (26.1)
  Satisfaction with breasts: number analyzed (Participants) | 95
  Satisfaction with breasts | 69 (20.7)

3. Secondary Outcome: Quality of Life as Measured by Breast-Q Questionnaire Scores at 24 Month Post-RT Timepoint
Description: as for outcome 2
Time Frame: 24 months post RT
Population: -80 sexual well-being subscale questionnaires were completed at this timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 90
score on a scale
  Physical well-being | 77.9 (23.1)
  Psychosocial well-being | 79.6 (22.4)
  Sexual well-being: number analyzed (Participants) | 80
  Sexual well-being | 63 (28.2)
  Satisfaction with breasts | 68.8 (21.6)

4. Secondary Outcome: Incidence of Acute and Late Radiation Complications Based on Common Terminology Criteria for Adverse Events (CTCAE) 4.0 Toxicity
Description: The proportion of patients with acute or late radiation complications, will be estimated. Any event longer than 3 months will be considered a late effect.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-05

5. Secondary Outcome: Local and Local Regional Recurrence Rate
Description: We will report the incidence of recurrence
Time Frame: Up to 60 months
Reporting Status: Not Posted, anticipated posting 2026-04

6. Secondary Outcome: Cost-effectiveness (CE) of Hypofractionated Radiation Versus Standard Fractionation
Description: Will be explored using cost data and quality adjusted life years (QALYs)
Time Frame: Up to 3 years
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 4/102
Other Adverse Events (participants affected / at risk) | 102/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=102)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Dysphasia (Gastrointestinal disorders) | 1 (2)
Myasthenia Gravis (Immune system disorders) | 1 (1)
Breast infection (Infections and infestations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=102)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 3 (3)
Eye disorders - Other, specify (Eye disorders) | 3 (4)
Eye pain (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 10 (11)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 7 (8)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 20 (23)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (7)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 3 (3)
Edema trunk (General disorders) | 3 (3)
Fatigue (General disorders) | 83 (112)
Fever (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 3 (5)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3)
Irritability (General disorders) | 3 (3)
Localized edema (General disorders) | 14 (17)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 14 (16)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 3 (3)
Autoimmune disorder (Immune system disorders) | 2 (2)
Bladder infection (Infections and infestations) | 1 (1)
Breast infection (Infections and infestations) | 1 (9)
Bronchial infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Nail infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 12 (12)
Urinary tract infection (Infections and infestations) | 9 (11)
Vaginal infection (Infections and infestations) | 4 (5)
Wound infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 90 (111)
Fall (Injury, poisoning and procedural complications) | 8 (10)
Fracture (Injury, poisoning and procedural complications) | 10 (10)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2 (2)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 5 (5)
Lymphocyte count decreased (Investigations) | 2 (2)
Weight gain (Investigations) | 4 (4)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (19)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (12)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 12 (13)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 22 (26)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (30)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 27 (27)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (18)
Cognitive disturbance (Nervous system disorders) | 2 (2)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 14 (17)
Hypersomnia (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 5 (5)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 6 (6)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Tremor (Nervous system disorders) | 4 (4)
Agitation (Psychiatric disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 5 (6)
Depression (Psychiatric disorders) | 8 (9)
Insomnia (Psychiatric disorders) | 12 (13)
Personality change (Psychiatric disorders) | 2 (2)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (3)
Restlessness (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Breast atrophy (Reproductive system and breast disorders) | 7 (7)
Breast pain (Reproductive system and breast disorders) | 65 (80)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 26 (31)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3)
Vaginal dryness (Reproductive system and breast disorders) | 5 (6)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (4)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (21)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 19 (20)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 65 (67)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 (3)
Menopause (Social circumstances) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 10 (15)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 39 (44)
Hypertension (Vascular disorders) | 4 (4)
Lymphedema (Vascular disorders) | 6 (6)
Thromboembolic event (Vascular disorders) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03345420/Prot_SAP_002.pdf
  • Informed Consent Form (2023-04-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03345420/ICF_001.pdf